CLINICAL TRIAL: NCT06621095
Title: Anlotinib Plus Benmelstobart and AG Versus AG in First-line Treatment of Advanced Metastatic Pancreatic Cancer: a Prospective, Randomized Controlled Clinical Trial (ALTER-PA-001)
Brief Title: Anlotinib Plus Benmelstobart and AG in First-line Treatment of Advanced Metastatic Pancreatic Cancer (ALTER-PA-001)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, liwei wang, Director of department of oncology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY2024-195-B
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer; First-line; Metastatic Pancreatic Cancer
Keywords: Metastatic Pancreatic Cancer; First-line; Immunotherapy; Angiogenesis inhibitors; Anlotinib
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — anlotinib; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anlotinib + benmelstobart + nab-paclitaxel + gemcitabine (Experimental): Initial treatment: anlotinib + benmelstobart + nab-paclitaxel + gemcitabine. Maintenance treatment (after 8 cycles): anlotinib + benmelstobart + gemcitabine.
  Interventions: Drug: anlotinib + benmelstobart + nab-paclitaxel + gemcitabine
- nab-paclitaxel + gemcitabine (Active Comparator): Initial treatment: nab-paclitaxel + gemcitabine. Maintenance treatment (after 8 cycles): gemcitabine.
  Interventions: Drug: nab-paclitaxel + gemcitabine

INTERVENTIONS:
Drug: anlotinib + benmelstobart + nab-paclitaxel + gemcitabine — 1. Before 8 cycles, anlotinib 8mg, po.qd, d1-14; benmelstobart: 1200mg, I.V., D1, Q3W; nab-paclitaxel: 125mg/m2, I.V., D1, D8, Q3W; gemcitabine: 1000/m2, ivgtt for more than 30min, D1, D8, Q3W. The above schemes are repeated every three weeks.
  2. After 8 cycles, the regimen is changed to anlotinib 8mg, po.qd, d1-14; benmelstobart: 1200mg, I.V., D1, Q3W; gemcitabine: 1000/m2, ivgtt for more than 30min, D1, D8, Q3W. The regimen is repeated every 3 weeks until the disease progresses or unacceptable toxicity.
  Arms: anlotinib + benmelstobart + nab-paclitaxel + gemcitabine
Drug: nab-paclitaxel + gemcitabine — 1. Before 8 cycles, nab-paclitaxel: 125mg/m2, I.V., D1, D8, Q3W; gemcitabine: 1000/m2, ivgtt for more than 30min, D1, D8, Q3W. The above schemes are repeated every three weeks.
  2. After 8 cycles, the regimen is changed to gemcitabine: 1000/m2, ivgtt for more than 30min, D1, D8, Q3W. The regimen is repeated every 3 weeks until the disease progresses or unacceptable toxicity.
  Arms: nab-paclitaxel + gemcitabine

SUMMARY:
This study is designed to explore the efficacy and safety of anlotinib combined with benmelstobart and AG (nab-paclitaxel and gemcitabine) as first-line treatment compared with AG (nab-paclitaxel and gemcitabine) in metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This is an open-label, multicenter, randomized controlled clinical trial. We plan to recruit 104 subjects and randomly assign them in a 2:1 ratio to either the experimental group receiving Anlotinib plus Benmelstobart plus Gemcitabine and Nab-Paclitaxel, or the control group receiving Gemcitabine and Nab-Paclitaxel as initial treatment. Each cycle of the aforementioned drugs will last three weeks, with tumor efficacy assessments conducted at the end of cycles 2, 4, 6, and 8. After 8 cycles of treatment, patients in the experimental group who achieve complete response (CR), partial response (PR), or stable disease (SD) will continue with maintenance therapy using Anlotinib plus Benmelstobart plus Gemcitabine. Similarly, after 8 cycles of treatment, patients in the control group who achieve CR, PR, or SD will continue with maintenance therapy using Gemcitabine monotherapy. Efficacy will be evaluated every 3 cycles (9 weeks) during the maintenance phase until disease progression or intolerability. This study aims to evaluate the efficacy and safety of the combination of Anlotinib and Benmelstobart with Gemcitabine and Nab-Paclitaxel in treating metastatic pancreatic cancer, providing a new treatment option for first-line therapy in patients with advanced metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old (including 18 and 75 years old);
* Histologically or cytologically confirmed diagnosis of metastatic pancreatic cancer;
* No prior systemic therapy for metastatic pancreatic cancer (allowable circumstances for inclusion include recurrence more than 6 months after neoadjuvant (chemo)radiotherapy plus radical surgery, or recurrence more than 6 months after the completion of adjuvant (chemo)radiotherapy or radical concurrent chemoradiotherapy);
* At least one measurable lesion according to RECIST v1.1 criteria (any previous radiotherapy-treated lesion that has not progressed cannot be selected as the target lesion);
* Eastern Cooperation Oncology Group (ECOG) performance status of 0-1;
* Life expectancy ≥ 3 months;
* Adequate organ and bone marrow function, meeting the following criteria (within 7 days before enrollment):

  1. Hematology:

     Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L Platelet count (PLT) ≥ 90 x 10^9/L Hemoglobin (HB) ≥ 90 g/L
  2. Biochemistry:

     Without liver metastasis: Serum total bilirubin (TBIL) ≤ 1.5x the upper limit of normal (ULN); with liver metastasis: TBIL ≤ 2.5 x ULN.

     Without liver metastasis: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN; with liver metastasis: ALT and AST ≤ 5 x ULN.

     Serum creatinine ≤ 1.5 x ULN and creatinine clearance rate ≥ 60 mL/min (calculated by the Cockcroft-Gault formula).
  3. Adequate coagulation function, defined as an international normalized ratio (INR) or a partial thromboplastin time (APTT) ≤ 1.5 x ULN.
* Women of childbearing age need to take effective contraceptive measures.

Exclusion Criteria:

* Previously received treatment with vascular endothelial growth factor receptor (VEGFR) inhibitors or immune checkpoint inhibitors;
* Received other systemic antitumor treatments within 4 weeks prior to enrollment, including chemotherapy, signal transduction inhibitors, hormone therapy, biological immunotherapy, targeted therapy, photodynamic therapy, and traditional Chinese medicine with clear antitumor indications;
* Have other untreated or concurrent malignancies (excluding cervical carcinoma in situ, well-controlled basal cell or squamous cell carcinoma of the skin, or malignancy that has been treated and has shown no signs or evidence of recurrence for more than 3 years, and patients who do not require systemic therapy at the time of signing informed consent);
* Presence of central nervous system (CNS) metastases or brain metastases before enrollment;
* Underwent any surgery (excluding biopsy), invasive treatment or operation without complete healing of surgical incisions within 4 weeks before enrollment (excluding venous catheter placement and puncture drainage);
* Received radiotherapy within 4 weeks before enrollment (allowable if at least 2 weeks have passed since palliative radiotherapy for bone lesions was completed before starting study medication);
* Previously received any organ transplantation;
* Clinically symptomatic ascites, pleural effusion, or pericardial effusion requiring puncture or drainage, or received drainage of effusions within 14 days before the first dose;
* International normalized ratio (INR) > 1.5 or partial thromboplastin time (APTT) > 1.5 x ULN;
* Clinically significant electrolyte abnormalities as determined by the investigator;
* Presence of active gastrointestinal diseases like active gastric and duodenal ulcers, ulcerative colitis, or unremoved tumors with active bleeding, or other conditions judged by the investigator to possibly cause gastrointestinal bleeding or perforation;
* Evidence or history of significant bleeding tendency or episodes within 3 months before enrollment (bleeding >30 mL, hematemesis, melena, or hematochezia), hemoptysis (> 5 mL of fresh blood within 4 weeks), or thromboembolic events such as stroke and/or transient ischemic attack within 12 months;
* Any severe and/or uncontrollable disease, including:

  1. History or presence of interstitial lung disease, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, severely impaired lung function, or other conditions that may interfere with the detection and management of suspected drug-related pulmonary toxicity.
  2. Clinically significant history of liver diseases, including active hepatitis (Hepatitis B reference: HBsAg positive with HBV DNA > 1 x 10^4 copies/mL or > 2000 IU/mL; Hepatitis C reference: HCV antibody positive with HCV RNA > 1 x 10^3 copies/mL), or other hepatitis, clinically significant moderate to severe hepatic cirrhosis; Note: Participants with eligible Hepatitis B or C must receive continuous antiviral treatment to prevent viral reactivation.
  3. Human immunodeficiency virus (HIV) antibody positivity.
  4. Uncontrolled hypertension (defined as systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg not controlled by medications);
  5. Poorly controlled cardiovascular clinical symptoms or diseases, including but not limited to acute myocardial infarction, malignant arrhythmias (including QTc > 450 ms for males and > 470 ms for females), ≥ Grade II congestive heart failure (New York Heart Association (NYHA) classification), or clinically significant abnormal myocardial enzyme levels as determined by the investigator;
  6. Active or uncontrollable severe infections (≥ NCI-CTC AE Grade 2 infections);
  7. Poorly controlled diabetes (fasting blood glucose (FBG) > 10 mmol/L);
  8. Proteinuria ≥ ++ on urinalysis and confirmed 24-hour urinary protein > 1.0 g;
  9. History or presence of autoimmune diseases, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener's granulomatosis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, autoimmune hepatitis, systemic sclerosis, Hashimoto's thyroiditis, autoimmune vasculitis, or autoimmune neuropathies (e.g., Guillain-Barre syndrome). Exceptions include stable hypothyroidism requiring hormone replacement therapy (including hypothyroidism due to autoimmune thyroid disease), psoriasis or vitiligo not requiring systemic treatment;
* Pregnant or breastfeeding women;
* Known history of allergy to investigational drug components;
* Participation in other clinical trials and treatment with investigational drugs within 4 weeks before enrollment;
* Any disease or condition that affects drug absorption or the inability of participants to take oral medications;
* Any other conditions judged by the investigator to be unsuitable for enrollment, including diseases, metabolic disorders, abnormal physical examination, laboratory result abnormalities, or any other conditions affecting the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 24 months
  The proportion of patients with complete response or partial response, using RESIST v1.1

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months
  Time from first-dose to the first documented disease progression or death
Disease Control Rate (DCR) | Up to 24 months
  The proportion of patients with complete response, partial response or stable disease, using RESIST v1.1
Duration of Response (DoR) | Up to 24 months
  Duration of response according to RECIST v1.1 (Response was assessed with CT or MRI using RECIST v1.1, Duration of response (DoR): DoR will only be performed in subjects who have a confirmed tumor response (CR or PR) after treatment
Overall Survival (OS) | Up to 24 months
  Overall Survival (OS) is defined as the time from enrollment to death from any cause.
Safety and tolerability by incidence, severity and outcome of adverse events | Until 30 day safety follow-up visit
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Wang, M.D., Principal Investigator — RenJi Hospital
Locations (1):
- Renji hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No